CLINICAL TRIAL: NCT00896142
Title: Optima CAD (Optimal Mechanical Evaluation)
Brief Title: Optima Coronary Artery Disease (CAD) (Optimal Mechanical Evaluation)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 0601112
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Heart Failure; Ischemic Cardiomyopathy
Keywords: ischemic cardiomyopathy; cardiac resynchronization therapy; LV structure and function
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To evaluate the impact of left ventricular (LV) lead location on LV mechanical function.

ELIGIBILITY:
Inclusion Criteria

1. Ischemic Cardiomyopathy
2. Left ventricular ejection fraction less than 40%
3. Clinical indication for invasive electrophysiology testing
4. Patient is at least 18 years of age

Exclusion Criteria

1. Unstable angina, acute myocardial infarction and/or revascularization procedure within 3 months
2. CVA or TIA within the past 6 months
3. Prosthetic heart valve
4. Patient is status post heart transplant
5. Women who are pregnant or with child -bearing potential and who are not on a reliable form of birth control. Women of child-bearing potential are routinely tested for pregnancy as part of the standard of care prior to EPS procedures being performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18+ years of age must be patients of UPMC Cardiovascular Institute
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: David S. Schwartzman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presybterian, Pittsburgh, Pennsylvania, United States